CLINICAL TRIAL: NCT05139147
Title: A Prospective, Multi-Center, Single Arm, Feasibility Study to Evaluate the DAISe Thrombectomy System During Neurointervention for Acute Ischemic Stroke; DAISe 1 Study
Brief Title: DAISe 1 Feasibility Study to Evaluate the DAISe Thrombectomy System for Acute Ischemic Stroke
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment/Recruitment
Sponsor: MIVI Neuroscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101995
Record Dates: First submitted 2021-11-09; First posted 2021-12-01 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DAISe Thrombectomy System (Experimental): Mechanical thrombectomy utilizing the DAISe Thrombectomy System, consisting of the DAISe Thrombectomy Device and DAISe Delivery Catheter, used with aspiration.
  Interventions: Device: DAISe Thrombectomy System

INTERVENTIONS:
Device: DAISe Thrombectomy System — DAISe Thrombectomy System for mechanical thrombectomy

SUMMARY:
The study is a prospective, multi-center, single arm, feasibility study that will enroll a maximum of 36 subjects. The maximum enrollment is 10 subjects per site. A maximum of 6 investigational centers in Europe will participate. Enrollment is expected to take about 9 months, subject participation will last about 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Pre-stroke (24 hours prior to stroke onset) independent functional status in activities of daily living with modified Rankin Score 0-1. Patient must be living in their own home, apartment or seniors lodge where no nursing care is required.
* Diagnosis of acute ischemic stroke and referred to interventional neuroradiology center for mechanical thrombectomy with study enrollment time planned within 8 hours from onset of symptoms.
* Disabling stroke defined as a baseline NIHSS > 6.
* Thrombolytic therapy (IV tPA) received within 4.5 hours of onset/ last known well according to prescribed dosing OR documented ineligibility for thrombolytic therapy.
* Confirmed symptomatic, large vessel occlusion of the intracranial internal carotid artery, middle cerebral artery, M1, or M2 with mTICI 0-1.
* The following baseline imaging criteria should be met: MRI criterion- volume of diffusion restriction visually assessed ≤50 mL OR ASPECTs score 5-10 or T criterion- ASPECTS 6-10 on imaging NE-CT, CTA and/or CTP available
* Signed informed consent from patient or legal representative or if applicable, documented medical necessity for inclusion in a clinical study in an emergency followed by signed informed consent.
* Patient is affiliated in the social security system.

Exclusion Criteria:

* Computed tomography (CT) or Magnetic Resonance Imaging (MRI) evidence of recent/ fresh hemorrhage on presentation.
* Clinical history, past imaging or clinical judgment suggests that the intracranial occlusion is chronic.
* Rapidly improving neurological deficits based on the investigator's clinical judgement.
* Pregnancy; if a woman is of child-bearing potential and urine or serum beta HCG test is positive.
* Severe contrast allergy or absolute contraindication to iodinated contrast.
* Renal failure (serum creatinine level ≥ 3 mg/dL or on dialysis).
* Severe, sustained hypertension resistant to treatment (SBP >185 mmHg or DBP >110 mmHg).
* Use of warfarin anticoagulation (or other applicable anti-vitamin k anticoagulants) with International Normalized Ratio (INR) > 3.0 at the time of the procedure or any known hemorrhagic or coagulation deficiency.
* Use of a direct thrombin inhibitor within the last 48 hours; partial thromboplastin time (PTT) > 2.0 times the normal prior to procedure.
* Cerebral vasculitis or evidence of active systemic infection.
* Suspicion of aortic dissection, presumed septic embolus or suspicion of bacterial endocarditis.
* Clinical symptoms suggestive of bilateral stroke or occlusions in multiple vascular territories (e.g., bilateral anterior circulation, or anterior/posterior circulation).
* Seizure due to stroke.
* Difficult endovascular access, difficult aortic arch or severe neurovascular tortuosity that will result in an inability to deliver endovascular therapy.
* Evidence of dissection in the carotid or target artery for treatment.
* Presence of a carotid artery stenosis or occlusion requiring balloon angioplasty or stenting at time of the procedure.
* A severe or fatal comorbid illness that will prevent improvement or follow-up or that will render the procedure unlikely to benefit the patient.
* Patient cannot undergo an MRI of the head due to MRI contraindication.
* Patient is unable or unwilling complete follow up visits.
* If before the stroke, the patient is under a legal protective measure, they will not be able to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-08-04 (Actual)

PRIMARY OUTCOMES:
Rate of first pass revascularization success | procedure
  First pass successful revascularization defined as mTICI (modified Treatment in Cerebral Ischemia) 2b-3 flow in the target vessel post-treatment with the DAISe Thrombectomy System used with aspiration.
Rate of symptomatic intracranial hemorrhage | 12-36 hours
  Symptomatic intracranial haemorrhage at 24 (+/-12) hours post-procedure as detected by CT/MRI with clinical deterioration of an NIHSS change of greater than or equal to 4

SECONDARY OUTCOMES:
Rate of successful revascularization with the DAISe Device | Procedure
  Successful revascularization of mTICI 2c-3 as a result of the first attempt with the DAISe Thrombectomy Device
Rate of procedural final successful revascularization | Procedure
  Successful revascularization of final mTICI 2b-3 at the end of the procedure
Rate of successful revascularization at procedure end | Procedure
  Successful revascularization of final mTICI 2c-3 at the end of the procedure
Rate of successful device use | Procedure
  Measured by the successful delivery and placement of the DAISe Device in the target artery
Procedure time | Procedure
  Time from groin puncture to successful revascularization defined as final mTICI 2b-3 flow
Complications | Procedure
  Rate of procedure and/or device related complications
Rate of ENT | Procedure
  Rate of embolization to a new vascular territory (ENT) during procedure
Infarct volume | 12-36 hours
  Infarct volume in MRI (FLAIR/Diffusion Weighted Imaging [DWI] combined)
Emboli | 12-36 hours
  Number of emboli outside of main infarct affected territory and outside the affected territory in high-resolution DWI
Intracranial hemorrhage | 12-36 hours
  Occurrence of all intracranial hemorrhage using the Heidelberg Bleeding Classification
Good functional outcome | 3 months
  Good functional outcome measured by Modified Rankin Score (measured 0 completely functional to 6 deceased) of 0-2
Mortality Rate | 3 months
  All cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Cognard, MD, PhD, Principal Investigator — University Hospital, Toulouse
Locations (6):
- France (6):
  - CHU Pellegrin, Bordeaux
  - CHU Montpellier, Montpellier
  - CHU Urbains, Nancy
  - CHU Bicetre Paris, Paris
  - Groupe Hospitalier Pitie-Salpetriere, Paris
  - Hôpital Purpan, Toulouse

IPD SHARING:
Plan to Share IPD: No